CLINICAL TRIAL: NCT05078138
Title: Impact of Erythropoietin on Hematological Adaptations and Physical Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-01H
Record Dates: First submitted 2021-08-06; First posted 2021-10-14 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Exercise-Induced Anemia; Physical Performance
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: Longitudinal study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exogenous Erythropoietin (Experimental): Recombinant human Erythropoietin subcutaneous injection of 50 IU/kg body mass 3 times per week for 4 week
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa — Subcutaneous injection of Epoetin Alfa 3 times per week for 4 weeks

SUMMARY:
Negative hematological adaptations due to prolonged periods of strenuous physical activity may, in part, contribute to declines in physical performance during military operations. Exogenous erythropoietin (EPO) is a potential intervention that may be used to maintain hemoglobin (hgb), hematocrit (Hct), and physical performance during periods of high physical activity. The objective of the current study is to determine the ability of EPO to maintain hgb, Hct, and physical performance compared to baseline measures. Additionally, EPO may result in non-hematological adaptations which increase mitochondria biogenesis and alter substrate oxidation. As such, this study will also assess the influence of EPO on whole-body and skeletal muscle substrate oxidation. Eight healthy physically active individuals will be recruited to participate in this longitudinal trial. After exercise practice sessions, volunteers will complete baseline physical performance (time trial) and substrate oxidation testing. Participants will then receive EPO injections 3 times per week for 4 weeks. Diet and exercise will be controlled during the injection period. Participants will undergo four weeks of an intense physical training exercise program. Every seventh day during the injection period a safety blood sample, assessing hematocrit, will be drawn, and participants will complete a 5 km time trial to determine the time course of changes in physical performance can be detected. After the 4 weeks of EPO injections volunteers will complete the same physical performance and substrate oxidation testing. Substrate oxidation will be assessed during 90-min steady-state load carriage (30% body mass) exercise on a treadmill at 55 ± 5% of VO2peak. 6-6-[2H2] glucose tracer technique and indirect calorimetry will be used measure substrate oxidation. Muscle biopsies will be performed to measure muscle glycogen, enzyme activity, and molecular markers of metabolism and inflammation before, and immediately and 3-hrs post exercise. Multiple blood samples will be collected throughout the study to determine alterations in hemoglobin, hematocrit, and markers of substrate metabolism, and inflammation. All study procedures will occur at USARIEM. The primary risks associated with this study include those associated with EPO injection, exercise, blood draws, and muscle biopsies.

DETAILED DESCRIPTION:
Healthy physically active individuals will be recruited to participate in this longitudinal trial. After baseline assessments of body composition, resting metabolic rate (RMR), VO2peak and exercise familiarization; volunteers will complete physical performance and substrate oxidation testing. Physical performance will be assessed using time trial. Substrate oxidation will be assessed by volunteers performing 90-min of steady-state load carriage (30% body mass) exercise on a treadmill at 55 ± 5% of their VO2peak. 6-6-[2H2] glucose will be used as a tracer to assess glucose turnover. Indirect calorimetry will be used to determine carbohydrate and fat oxidation. Muscle biopsies will be performed to measure muscle glycogen, enzyme activity, and molecular markers of substrate metabolism before, immediately after, and 3-hrs post exercise. Multiple blood samples will be collected on substrate oxidation protocol days. To minimize carry over effects of muscle biopsies on subsequent exercise performance, volunteers will not exercise for 3 days. During the first two days of this period, volunteers will undergo carbon monoxide (CO) rebreathing to measure Hgb mass and blood volume. Volunteers will then receive EPO injections 3 times a week for 4 weeks. During the injection period all volunteers will have safety blood draws to assess Hct once a week. Volunteers will also complete a physical performance test once a week to determine time course change in performance with EPO compared to baseline. Exercise training will be controlled during the injection phase, consisting of a combination of endurance- and resistance-type exercise. During the final week of the injection phase body composition, resting metabolic rate (RMR) and VO2peak will be reassessed. At the end of the 4-week injection phase volunteers will complete a final physical performance test and substrate oxidation protocol, followed by two CO rebreathing tests on subsequent days. All food and beverages (except water) will be provided to volunteers beginning at the pre injection physical performance and substrate oxidation through the duration of the study. All data collection will occur at USARIEM.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years
* Weight stable (±5 lbs) for at least 2 months prior to the start of the study
* Body mass index (BMI) between 18.5-30 kg/m2
* Recreationally active (minimum 2-4 days per week aerobic and/or resistance exercise)
* Refrain from taking any NSAIDS (i.e., aspirin, Advil®, Aleve®, Naprosyn®, or any aspirin-containing product for 10 days before and at least 5 days AFTER each muscle biopsy. (*Tylenol® or acetaminophen is ok to use if needed for discomfort)
* Refrain from the use of alcohol and nicotine while on study diets
* Supervisor approval for federal civilian employees working within the US Army Natick Soldier Systems Center

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (i.e., kidney disease, diabetes, cardiovascular disease, hypertension etc.)
* Personnel or family history of blood clots
* Disease or medication (i.e., diabetes medications, statins, corticosteroids, etc) that affects macronutrient utilization and/or the ability to participate in strenuous exercise
* Allergies or intolerance to foods (including but not limited to lactose intolerance/milk allergy), vegetarian practices, or medications (including, but not limited to, lidocaine or phenylalanine) to be utilized in the study
* History of inflammatory bowel disease
* History of seizures
* Anemia (HCT < 38) and Sickle Cell Anemia/Trait
* Abnormal PT/PTT test or problems with blood clotting
* Present condition of alcoholism, use of nutritional/sports supplements, anabolic steroids, or other substance abuse issues
* History of malignancy
* Use of oral contraceptives or hormone replacement therapy due to increased risk of clotting
* Musculoskeletal injuries that compromise the ability to exercise
* Blood donation within 8 weeks of beginning the study
* Are unwilling or unable to eat study diets and foods provided and/or follow exercise prescriptions
* Pregnancy, post-partum status, or breastfeeding

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exogenous Erythropoietin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exogenous Erythropoietin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 8
VO2peak [Mean (Standard Deviation); unit: ml/kg/min] | 44 (2)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Hemoglobin
Description: Determine the effects of EPO on hemoglobin concentration compared to baseline during 4 weeks of overtraining.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Exogenous Erythropoietin
Number analyzed (Participants) | 8
g/dL | 1.46 (0.71)

2. Primary Outcome: Time to Complete 5 km Time Trial
Description: Determine the time course change in time to complete a 5 km treadmill run with EPO compared to baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exogenous Erythropoietin
Number analyzed (Participants) | 8
seconds | -166 (143)

3. Secondary Outcome: Rate of Fat Oxidation
Description: Assess the influence of EPO non-hematological adaptation (carbohydrate and fat oxidation rates and skeletal muscle substrate oxidation and glucose turnover rates) following 4 weeks of overtraining compared to baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Exogenous Erythropoietin
Number analyzed (Participants) | 8
g/min | 0.08 (0.16)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Exogenous Erythropoietin
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT05078138/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT05078138/SAP_003.pdf
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT05078138/ICF_001.pdf